CLINICAL TRIAL: NCT00340158
Title: The Establishment of an Inflammatory Breast Cancer Registry and Biospecimen Repository
Brief Title: Establishing an Inflammatory Breast Cancer Registry
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903214; 03-C-N214
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Inflammatory Breast Cancer
Keywords: Mammary; Diagnosis; Aggressive; Pathology; Epidemiology
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Disease; Aggression

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Inflammatory breast carcinoma (IBC) is an extremely rare, aggressive form of breast cancer that disproportionately impacts young women. IBC often affects the skin of the breast, as well as the breast itself, making it appear inflamed. The purpose of this study is to collect data and information on IBC patients so that researchers can study factors associated with IBC. The data and information collected will be used to establish the IBC Registry, a private cancer registry.

Approximately 300 persons who are 18 years or older and who have been diagnosed with IBC will participate in this study. Participants will provide researchers with access to their medical and pathology records, slides, tissue, and x-rays. They also will consent to a 15-minute telephone interview concerning general information about themselves and the initial manifestation of IBC and to a 30-minute interview about their medical history.

DETAILED DESCRIPTION:
Inflammatory breast carcinoma (IBC) is an extremely rare, aggressive form of breast carcinoma that disproportionately affects young women. Clinical features of IBC include warmth, redness, edema, skin dimpling and rapid enlargement; the hallmark pathologically is dermal lymphatic invasion. Minimal criteria necessary for a clinical diagnosis of IBC have been debated and relatively little is known about the epidemiology, pathogenesis and molecular characteristics of these very lethal tumors. This project, funded by a grant from the Department of Defense awarded to PHL, would develop a national registry of approximately 300 volunteers (aged 18 years or older) with IBC. Subjects will provide access to medical records, pathology records, slides, blocks and tissue (fixed and frozen) and x-rays and consent to an interview. Recruitment will be performed at collaborating institutions and through an IBC research foundation (Owen Johnson) that maintains a website and e-mail contact lists. The registry resources would be made available collaboratively to anyone in the breast cancer research community, based on merit as determined by a designated committee. Central aims of the study include determining whether clinically or pathologically defined IBC differs in clinical behavior or biologically, identifying markers in IBC that may provide useful information about the aggressive potential of breast cancers generally, and evaluation of tissue for mouse mammary tumor virus (MMTV) related sequences. The purpose of this IRB submission is to review the role of MES as a collaborating pathologist on this study. Enrollment is closed as of this time.

ELIGIBILITY:
* Patients will be recruited from collaborating institutions throughout the US and through the IBC research foundation (established by patient advocate, Mr. Owen Johnson), which maintains a website and a research e-mail list. The goal is to recruit approximately 300 volunteers, at least 18 years of age or older.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Levine PH, Steinhorn SC, Ries LG, Aron JL. Inflammatory breast cancer: the experience of the surveillance, epidemiology, and end results (SEER) program. J Natl Cancer Inst. 1985 Feb;74(2):291-7. PMID 3856043
- [Background] Chang S, Parker SL, Pham T, Buzdar AU, Hursting SD. Inflammatory breast carcinoma incidence and survival: the surveillance, epidemiology, and end results program of the National Cancer Institute, 1975-1992. Cancer. 1998 Jun 15;82(12):2366-72. PMID 9635529
- [Background] Mourali N, Levine PH, Tabanne F, Belhassen S, Bahi J, Bennaceur M, Herberman RB. Rapidly progressing breast cancer (poussee evolutive) in Tunisia: studies on delayed hypersensitivity. Int J Cancer. 1978 Jul 15;22(1):1-3. doi: 10.1002/ijc.2910220102. PMID 681022